CLINICAL TRIAL: NCT03103945
Title: Prospective Physician-Initiated Observational Study of The Contact Detection System (CDS) in Patients Undergoing Radiofrequency Ablation Using the Niobe™ Remote Magnetic Navigation System (STAR)
Brief Title: Prospective Physician-Initiated Observational Study of The Contact Detection System (CDS) in Patients Undergoing Radiofrequency Ablation Using the Niobe™ Remote Magnetic Navigation System
Acronym: STAR
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Anne-Marie Noten, MD, Erasmus Medical Center
Other Study IDs: CLIN-022
Record Dates: First submitted 2017-03-26; First posted 2017-04-07 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation; Catheter Ablation
Keywords: Atrial Fibrillation; Atrial Arrhythmia; Arrhythmias, Cardiac; Cardiac Diseases; Electrophysiologic Techniques, Cardiac; Electrophysiology; Remote Magnetic Navigation; Contact Detection System
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cardiac arrhythmias undergoing RF ablation: Patients with cardiac arrhythmias will be undergoing RF ablation using the Niobe Remote Magnetic Navigation System with CDS as their standard of care. System performance data will only be collected during the RF ablation procedure. Outcome measures will be evaluated with the CDS connected and without the CDS connected within all patients.
  Interventions: Device: CDS box connection of the Niobe™ Remote Magnetic Navigation System

INTERVENTIONS:
Device: CDS box connection of the Niobe™ Remote Magnetic Navigation System — For all subjects included in the study, the ablation procedure will be started per standard of care. First mapping, pacing and electrocardiograms of the right atrium will be evaluated without the CDS box connected. Second the CDS box will be connected to the catheter and mapping, pacing and electrocardiograms will be recorded again. Next, ablation will be conducted per standard of care.

SUMMARY:
This observational study evaluates peri-procedural results of the Niobe™ Remote Magnetic Navigation (RMN) ES system using the contact detection system (CDS) in patients undergoing standard of care radiofrequency ablation of cardiac arrhythmias.

The objective of this observational study is to confirm system performance of the CDS and that it does not alter pacing, electrocardiograms, or mapping during RF ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical indication for RF ablation of cardiac arrhythmias with the Niobe Remote Magnetic Navigation system
* patients referred to one of the participating ablation centers
* written informed consent

Exclusion Criteria:

* presence of a atrial thrombus or left atrial appendage (LAA) thrombus seen on (contrast) echocardiography or MRI
* contra-indication for general anesthesia
* age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participant sampling of patients who will receive RF ablation of cardiac arrhythmias with the Niobe Remote Magnetic Navigation system.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Mapping quality | One day - during ablation procedure
  Physician's and technician's subjective score of the quality of mapping the right atrium without CDS box connected and with CDS box connected
Pacing thresholds | One day - during ablation procedure
  Pacing thresholds of three separate areas of the right atrium without CDS box connected and pacing thresholds of the same three areas with CDS box connected
Pacing capture | One day - during ablation procedure
  Pacing capture of three separate areas of the right atrium without CDS box connected and pacing capture of the same three areas with CDS box connected
Electrocardiograms | 10 months - ECGs will be evaluated after inclusion is completed
  Difference between and disturbance of the intracardiac electrocardiograms without the CDS box connected versus with the CDS box connected, evaluated by two independent and blinded electrophysiologists

SECONDARY OUTCOMES:
Number of procedure related major adverse events, attributed to the CDS system | 30 days
  Major adverse events: death, acute myocardial infarction (AMI) or coronary artery damage, major bleeding - type III and V, abdominal bleeding, tamponade > 80cm3, late tamponade, ischemic cerebral event
Number of procedure related minor adverse events, attributed to the CDS system | 30 days
  Minor adverse events: post procedural precordial pain, phrenic nerve injury, minor bleeding - type II
Number of acute procedure succes | 1 day - during ablation procedure
  Number of procedures with successful electrical isolation of ablated area

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands